CLINICAL TRIAL: NCT06856720
Title: Effects of Neuromuscular Electrical Stimulation and Aerobic and Resistance Exercise on Glycemic Control in Older Adults With Type 2 Diabetes
Brief Title: Impact of NMES, Aerobic, and Resistance Exercise on Glycemic Control in Older Adults With Type 2 Diabetes
Acronym: NMES4GliCon
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carlos Tavares (Other)
Collaborators: University of Salamanca (Other); Escola Superior de Tecnologia da Saúde de Coimbra (Other); Instituto Piaget (Other)
Responsible Party: Sponsor-Investigator, Carlos Tavares, Effects of Neuromuscular Electrical Stimulation and Aerobic and Resistance Exercise on Glycemic Control in Older Adults with Type 2 Diabetes: A Randomized Controlled Trial, University of Salamanca
Organization: University of Salamanca (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMES_T2DM_2025
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Glycemic Control; Neuromuscular Electrical Stimulation; Type 2 Diabetes Mellitus; Aerobic Exercise; Resistance Training; Elderly Population; Diabetes Management; Health Literacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial (RCT) with three arms: 1) Neuromuscular Electrical Stimulation (NMES) group, 2) Aerobic and Resistance Exercise group, and 3) Health Literacy Group. Participants will be randomized to one of the three groups and undergo interventions for 12 weeks, with initial, final, and follow-up assessments at 30, 60, and 90 days to evaluate the efficacy and maintenance of effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NMES Intervention Group (Experimental): Participants in this arm will receive neuromuscular electrical stimulation (NMES) for 30 minutes, three times per week, for 12 weeks. The sessions will be supervised by a physical therapist. NMES will be applied to large muscle groups, such as the quadriceps, using specific parameters (5 Hz frequency, 400 μs pulse duration, 4 seconds stimulation on, 12 seconds rest off), adjusted to the maximum tolerable intensity for each participant. This group aims to evaluate the effect of NMES on glycemic control and quality of life in older adults with type 2 diabetes mellitus (T2DM).
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES)
- Exercise Intervention Group (Experimental): Participants in this arm will engage in a combined aerobic and resistance exercise program three times per week for 12 weeks. The program will consist of 20 minutes of aerobic exercise (60-75% of maximum heart rate or moderate perceived effort) and 20 minutes of resistance training (50-70% of one-repetition maximum, focusing on large muscle groups). This exercise program will be supervised by a physical therapist and adapted to the participants' physical capabilities. This arm aims to compare the effects of exercise on glycemic control and quality of life in older adults with T2DM.
  Interventions: Behavioral: Aerobic and resistance exercise
- Health Education Group (Active Comparator): Participants in this arm will receive health education focused on diabetes management, including lifestyle changes and strategies for improving glycemic control. The sessions will be led by trained healthcare providers and will focus on diet, exercise, and self-management strategies. The goal is to assess the effects of health education on fasting glucose levels and quality of life in older adults with T2DM.
  Interventions: Behavioral: Health literacy education

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation (NMES) — Participants will receive NMES application for 30 minutes, three times a week, over a period of 12 weeks. The sessions will be supervised by a physiotherapist. Large muscle groups (quadriceps) will be used, with the following current parameters: frequency of 5 Hz, pulse width of 400 μs, 4 seconds of stimulation (on) for 12 seconds of rest (off), and intensity adjusted to the maximum tolerable level for the patient. These parameters are based on studies that have shown significant improvements in glycemic control and insulin sensitivity, especially in older adults with type 2 diabetes.
  Arms: NMES Intervention Group
Behavioral: Aerobic and resistance exercise — This group will participate in an exercise program combining aerobic and resistance activities, performed three times per week for 12 weeks. The activities will be adapted to the participants' physical capabilities and supervised by a physiotherapist. The program follows the international recommendations and it includes a 5-minute warm-up with flexibility exercises, 20 minutes of aerobic exercise at 60-75% of maximum heart rate or moderate perceived exertion, 20 minutes of resistance exercise at 50-70% of one-repetition maximum (1RM) focusing on large muscle groups (10-15 repetitions per exercise, 1-3 sets), and a 5-minute cool-down with static stretching and breathing exercises for relaxation.
  Arms: Exercise Intervention Group
Behavioral: Health literacy education — Participants will receive educational sessions on diabetes management, the role of exercise in glycemic control, and strategies to enhance adherence to physical activity.
  Arms: Health Education Group

SUMMARY:
This study aims to evaluate the effects of neuromuscular electrical stimulation (NMES), aerobic and resistance exercise, and health literacy intervention on fasting glucose levels and quality of life in older adults with type 2 diabetes (T2DM). Given the growing prevalence of T2DM in aging populations and the associated health risks, identifying effective interventions is crucial. The randomized controlled trial (RCT) will include participants aged 60+ with T2DM, randomly assigned to one of three groups: NMES, structured exercise, or a health literacy control group. Outcomes will be assessed at baseline, post-intervention (12 weeks), and follow-up (30, 60, and 90 days). The primary outcome is fasting glucose levels, while secondary outcomes include adherence, treatment satisfaction, and quality of life. This study seeks to provide evidence on alternative approaches for glycemic control in elderly individuals, particularly those with limited physical activity capacity.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) investigates the effects of neuromuscular electrical stimulation (NMES), aerobic and resistance exercise, and a health literacy program on glycemic control and quality of life in older adults with type 2 diabetes mellitus (T2DM). Given the increasing prevalence of T2DM among the elderly and the challenges associated with its management, this study aims to evaluate alternative, accessible interventions that may improve metabolic health and overall well-being.

Study Design:

A parallel-group, randomized controlled trial with three intervention arms:

NMES Group: Participants will undergo NMES sessions targeting large muscle groups (quadriceps) for 30 minutes, three times per week over a period of 12 weeks. The stimulation parameters will be adjusted based on tolerability, following evidence-based protocols for improving glucose uptake.

Exercise Group: Participants will engage in a structured exercise program combining aerobic and resistance training, performed three times per week for 12 weeks under professional supervision. The protocol will follow international guidelines for T2DM exercise interventions.

Health Literacy Group: Participants will receive educational sessions on T2DM management, including lifestyle modifications, dietary recommendations, and glucose monitoring strategies.

Primary Outcome:

- Fasting glucose levels (measured at baseline, post-intervention, and follow-up at 30, 60, and 90 days).

Secondary Outcomes:

* Adherence to the intervention;
* Treatment satisfaction;
* Quality of life (measured using the ADDQoL-18 questionnaire);
* Impact of baseline physical activity level and functional capacity on intervention response;

Significance:

This study will explore the potential of NMES as an alternative or adjunct therapy for older adults with limited physical activity capacity. By comparing NMES with traditional exercise and health education, it will provide valuable insights into the feasibility, effectiveness, and long-term sustainability of these interventions for glycemic control in elderly populations with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes Mellitus (T2DM).
* Aged 60 years or older.
* Sufficient cognitive ability to understand study instructions.
* Institutionalized in nursing homes or similar settings.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Severe cardiovascular diseases (e.g., heart failure, recent myocardial infarction).
* Musculoskeletal conditions that prevent exercise participation (e.g., severe arthritis, unhealed fractures).
* Intensive insulin therapy with high risk of hypoglycemia or significant glycemic control issues.
* Participation in other clinical trials that could interfere with this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Fasting Blood Glucose Levels | Baseline, after 12 weeks of intervention, and at follow-ups (30, 60, and 90 days post-intervention).
  Measurement of fasting blood glucose levels using standardized blood collection and analysis.
Glycemic Control (HbA1c) | Baseline, after 12 weeks of intervention, and at follow-ups (30, 60, and 90 days post-intervention).
  Measurement of hemoglobin A1c (HbA1c) levels using a blood test to assess long-term glycemic control.

SECONDARY OUTCOMES:
Health-Related Quality of Life | Baseline, after 12 weeks of intervention, and at follow-ups (30, 60, and 90 days post-intervention).
  Assessment of quality of life related to diabetes using the Audit of Diabetes Dependent Quality of Life - 18 (ADDQoL-18, Portuguese version) questionnaire. The ADDQoL-18 produces a weighted score ranging from -9 (worst possible quality of life) to +3 (best possible quality of life), with higher scores indicating better quality of life.questionnaire.
Treatment Adherence Rates | After 12 weeks of intervention.
  Percentage of participants who complete the intervention sessions (NMES, exercise, or health literacy), measured through session attendance records.
Participant Satisfaction | After 12 weeks of intervention.
  Measurement of participant satisfaction with the intervention using the Diabetes Treatment Satisfaction Questionnaire (DTSQ). The DTSQ produces a total score ranging from 0 (lowest satisfaction) to 36 (highest satisfaction), with higher scores indicating greater satisfaction with the treatment.

OTHER OUTCOMES:
Baseline Physical Activity Level | Baseline.
  Measurement of baseline physical activity level using a pedometer, expressed as the average daily step count recorded over 7 consecutive days. This measure will be used as a covariate in the analysis to adjust for potential baseline differences.
Baseline Physical Fitness Level | Baseline.
  Assessment of baseline physical fitness using the Senior Fitness Test (SFT), which includes multiple components (2-minute step test, chair stand test, arm curl test, chair sit-and-reach test and back scratch test). These measures will be used as covariates in the analysis to adjust for potential baseline differences.